CLINICAL TRIAL: NCT02420444
Title: A Phase I Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Safety and Immunogenicity of BCG and AERAS-404 Administered as a Prime-Boost Regimen to HIV-Negative, TB-Negative, BCG-Naive Adults
Brief Title: A Study for Safety and Immunogenicity of BCG and AERAS-404 in HIV-Negative, TB-Negative, BCG-Naive Adults
Acronym: C-013-404
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aeras (Other)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C-013-404
Record Dates: First submitted 2015-04-15; First posted 2015-04-17 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- BCG SSI prime with Placebo (Placebo Comparator): All subjects received BCG Vaccine SSI, 2-8 x 10^5 CFU (BCG) on Study Day -42.
  Placebo containing 0,8 mL sterile buffer consisting of 10 mmol Tris and 169 mmol NaCl aqueous solution was administered on Study Days 0, 56, and 231.
  Interventions: Biological: BCG SSI; Biological: Placebo
- BCG SSI prime with Placebo and AERAS-404 (Experimental): All subjects received BCG Vaccine SSI, 2-8 x 10^5 CFU (BCG) on Study Day -42.
  Placebo on Study Day 0 followed by AERAS-404 50/500 on Study Days 56 and 231.
  AERAS-404 50/500 was a fixed dose combination of H4 50 mcg and IC31 500 nmol (KLK equivalent). H4 and IC31 adjuvant were supplied as separate single-dose vials containing frozen product as follows:
  * H4 antigen: 500 mcg/mL (100 mcg/0.2 mL), in 10 mmol/L Tris-HCl, pH 8.3.
  * IC31 adjuvant: 1250 nmol/mL (1000 nmol/0.8 mL) KLK equivalent, in 10 mmol/L Tris-HCl and 169 mmol/L NaCl.
  Interventions: Biological: BCG SSI; Biological: Placebo; Biological: AERAS-404
- BCG SSI prime with AERAS-404 (Experimental): All subjects received BCG Vaccine SSI, 2-8 x 10^5 CFU (BCG) on Study Day -42.
  AERAS-404 50/500 on Study Days 0, 56, and 231.
  AERAS-404 50/500 was a fixed dose combination of H4 50 mcg and IC31 500 nmol (KLK equivalent). H4 and IC31 adjuvant were supplied as separate single-dose vials containing frozen product as follows:
  * H4 antigen: 500 mcg/mL (100 mcg/0.2 mL), in 10 mmol/L Tris-HCl, pH 8.3.
  * IC31 adjuvant: 1250 nmol/mL (1000 nmol/0.8 mL) KLK equivalent, in 10 mmol/L Tris-HCl and 169 mmol/L NaCl.
  Interventions: Biological: BCG SSI; Biological: AERAS-404

INTERVENTIONS:
Biological: BCG SSI — The dose volume administered for BCG was 0.1 mL, and the mode of administration was ID injection to the deltoid area.
  Other Names: BCG Vaccine SSI Danish; bacillus Calmette-Guérin
Biological: Placebo — This is the identical buffer solution in which H4:IC31 was formulated. The dose volume administered for Placebo was 0.5mL, and the mode of administration was an IM injection.
  Other Names: Sterile buffered saline
  Arms: BCG SSI prime with Placebo; BCG SSI prime with Placebo and AERAS-404
Biological: AERAS-404 — AERAS-404 vaccine was reconstituted on site by adding 0.2 mL H4 antigen solution to 0.8 mL IC31 adjuvant solution. The dose volume administered for AERAS-404 was 0.5mL, and the mode of administration was an IM injection.
  Other Names: H4:IC31
  Arms: BCG SSI prime with AERAS-404; BCG SSI prime with Placebo and AERAS-404

SUMMARY:
70 subjects received BCG intradermally at Study Day -42, then at Study Day 0 were randomized to receive AERAS-404 50 mcg H4/500 nmol IC31 intramuscularly as a 3-dose (N=30) or 2-dose (N=30) regimen, or placebo (N=10). Subjects were vaccinated on Study Days 0, 56, and 231, and followed through Study Day 259.

DETAILED DESCRIPTION:
A total of 70 subjects who had received BCG at Study Day -42 were randomized on Study Day 0 to receive 3 doses of placebo (N=10); 1 dose of placebo followed by 2 doses of AERAS-404 (N=30; AERAS-404 2 dose regimen); or 3 doses of AERAS-404 (N=30; AERAS-404 3 dose regimen). A total of 69 (98.6%) subjects completed the study; the remaining subject, in the AERAS-404 2 dose regimen, withdrew consent. All 70 subjects received the first and second vaccinations with placebo or AERAS-404 on Study Days 0 and 56, and 67 (95.7%) subjects received the third vaccination on Study Day 231. Three subjects did not receive the Study Day 231 vaccination (2 in the AERAS-404 2 dose regimen, 1 due to withdrawal of consent and 1 due to pregnancy [the subject delivered a healthy boy without complications and was followed to study completion]; and 1 in the AERAS-404 3 dose regimen, due to inability to discontinue daily isotretinoin started after the second vaccination [the subject was followed to study completion]).

ELIGIBILITY:
Inclusion Criteria:

1. Had completed the written informed consent process.
2. Was male or female.
3. Was age ≥ 18 years and ≤ 50 years.
4. Agreed to stay in contact with the study site for the duration of the study, provide updated contact information as necessary, and had no current plans to move from the study area for the duration of the study.
5. Agreed to avoid elective surgery for the duration of the study.
6. Had completed simultaneous enrollment in Aeras Vaccine Development Registry protocol.
7. For female subjects: agreed to avoid pregnancy from 28 days prior to Study Day 0 through the duration of the study.
8. Had general good health, confirmed by medical history and physical examination.
9. Had body mass index (BMI) between 18 and 33 (weight/height2) by nomogram.

Exclusion Criteria:

1. Oral temperature ≥37.5°C.
2. Abnormal CBC laboratory values (per local laboratory parameters) from blood collected at screening (>5% above ULN or >5% below LLN).
3. Abnormally elevated laboratory values (per local laboratory parameters) from blood collected at screening for ALT, AST, GGT, total bilirubin, alkaline phosphatase (ALP), blood urea nitrogen (BUN), creatinine, prothrombin time (PT), or partial thromboplastin time (PTT) (>10% above ULN).
4. Abnormal urinalysis that, in the opinion of the investigator, was clinically significant.
5. Positive screening urine test for illicit drugs (opiates, cocaine, amphetamines).
6. History or evidence of active or latent tuberculosis infection, including a positive QuantiFERON-TB test, a history of a positive TST, or abnormal chest X-ray findings that in the opinion of the investigator were evidence of tuberculosis.
7. Residence longer than 6 months in a high-burden country (per WHO 2010 TB Report).
8. Shared a residence within 1 year prior to Study Day -42 with an individual on anti-tuberculosis treatment or with culture- or smear-positive pulmonary tuberculosis.
9. Previous treatment for active or latent tuberculosis infection.
10. History or evidence of autoimmune disease.
11. History or evidence of any past, present, or future possible immunodeficiency state, including laboratory evidence of HIV 1 infection.
12. History or evidence of chronic hepatitis, including hepatitis B core antibody or hepatitis C antibody.
13. Received a TST within 90 days prior to Study Day -42.
14. Received a systemic antibiotic with 14 days prior to Study Day -42.
15. Received BCG vaccination or BCG immunotherapy prior to Study Day -42.
16. Received investigational Mtb vaccine.
17. Participation in any other investigational study during the study period.
18. Current household contact with an individual with known significant immunosuppression.
19. Occupational exposure that would have put an immunocompromised individual at risk, unless measures could be taken to reduce this risk to an acceptable level (e.g., plaster on the injection site).
20. Received immunoglobulin or blood products within 90 days prior to Study Day -42.
21. Received any investigational drug therapy or investigational vaccine within 180 days prior to Study Day -42.
22. Received any licensed vaccine within 45 days prior to Study Day -42 (note: the use of licensed vaccines medically indicated during the study was permitted at any time).
23. Received immunosuppressive medications other than inhaled or topical immunosuppressants within 45 days prior to Study Day -42.
24. Inability to discontinue daily medications other than the following during the study: oral contraceptives, vitamins, nonprescription nutritional supplements, aspirin, antihistamines, antihypertensives, antidepressants.
25. All female subjects: currently pregnant or lactating/nursing; positive screening urine pregnancy test; or positive urine pregnancy test on the day of any study vaccination.
26. History or evidence of allergic disease or reaction that, in the opinion of the investigator, may have compromised the safety of the subject.
27. History or evidence of dermatologic disease that, in the opinion of the investigator, may have interfered with the assessment of injection site reactions.
28. History or evidence of any other acute or chronic disease that, in the opinion of the investigator, may have interfered with the evaluation of the safety or immunogenicity of the vaccine or compromise the safety of the subject.
29. Medical, psychiatric, occupational, or substance abuse problems that, in the opinion of the investigator, would make it unlikely that the subject would comply with the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Number of unsolicited, solicited, and serious adverse events (SAEs). | 259 days
  Includes injection site AEs and systemic AEs.

SECONDARY OUTCOMES:
Immunogenicity of BCG and a 2- or 3-dose regimen of AERAS-404 measured by intracellular staining assay (ICS). | 259 Days
  ICS permits the detection of antigen-specific cytokine responses with a distinction between CD4+ and CD8+ T cells.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Pantaleo, MD, Principal Investigator — Centre Hosptialier Universitaire Vaudois (CHUV)
Locations (1):
- Centre Hosptialier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided